CLINICAL TRIAL: NCT06436040
Title: A Mechanism Study to Investigate the Difference in Efficacy of Neoadjuvant PD-1 Blockade Combined With Chemotherapy in the Treatment of IIA-IIIB Stage Lung Squamous Cell Carcinoma
Brief Title: Mechanism Study to Investigate Difference in Efficacy of Neoadjuvant Chemoimmunotherapy in Lung Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202311-10
Record Dates: First submitted 2024-01-22; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Tumor Microenvironment; Lung Squamous Cell Carcinoma; Neoadjuvant Chemoimmunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — pre-treatment and post-treatment tumors from patients with operable locally advanced lung squamous cell carcinoma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MPR(major pathological response): defned as having no more than 10% residual viable tumor cells by routine hematoxylin and eosin (H&E) staining after therapy
  Interventions: Other: Pathological response assessment
- non-MPR: defned as having more than 10% residual viable tumor cells by routine hematoxylin and eosin (H&E) staining after therapy
  Interventions: Other: Pathological response assessment

INTERVENTIONS:
Other: Pathological response assessment — The pathological response classification in our study was based on the histopathologic examination of the surgically resected specimens reviewed by two experienced pathologists.

SUMMARY:
To explore mechanisms of immunotherapy resistance and relation to changes in the TME before and after PD-1 blockade combined with chemotherapy

DETAILED DESCRIPTION:
The biobank of thoracic surgery department of Tangdu Hospital collected pre-treatment tissues from patients during endoscopy. The investigators retrospectively summarized the clinical characteristics of these patients and patients with operable locally advanced lung squamous cell carcinoma were selected and followed.

The investigators plan to employ snRNA-seq and scRNA-seq respectively to profile 20 samples of paired pre-treatment and post-treatment tumors from ten patients (discovery cohort) to create a cell atlas for analysis, and spatial transcriptomics to examine 8 samples from four patients. In discovery cohort, estimated 5 patients achieve major pathological response (MPR) and 5 patients achieve non-MPR after NICB.

After analyzing the results of discovery cohort, the investigators will collect frozen tissues and formalin-fixed, paraffin-embedded (FFPE) tissue from our biobank for bulk RNA-seq analysis or immunohistochemistry (IHC) staining as validation cohort to further investigate the predictive value and biological significance of our markers.

ELIGIBILITY:
Inclusion Criteria:

1. aged 40 to 80 years;
2. had histologically confirmed LUSC with operable locally advanced stage
3. no prior anti-tumor therapy; received neoadjuvant immunotherapy consisting of three cycles of anti-PD-1 ICB plus nab-paclitaxel and carboplatin
4. pre-treatment tissues

Exclusion Criteria:

1. the presence of central nervous system metastases
2. the presence of immunodeficiency disease; previous therapies with immunosuppressants within 14 days prior to the initiation of study treatment;
3. uncontrolled hypertension
4. history of or having pulmonary fibrosis or interstitial lung disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients enrolled in this study had histologically confirmed LUSC with operable locally advanced stage, no prior anti-tumor therapy, and received neoadjuvant immunotherapy consisting of three cycles of anti-PD-1 ICB plus nab-paclitaxel and carboplatin
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-11-16 (Estimated); Study Completion 2025-05-16 (Estimated)

PRIMARY OUTCOMES:
Pathological response assessment | through study completion, an average of 2 year
  MPR: Resected tumors with ≤10% viable tumor cells were considered to have a MPR

CONTACTS AND LOCATIONS:
Locations (1):
- Hongtao Duan, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No